CLINICAL TRIAL: NCT00442481
Title: Escitalopram and Sleep Architecture in Patients With Major Depressive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Lundbeck Israel (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-06-4205-JL-CTIL
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-03

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Escitalopram; Cipralex; Sleep; REM; SWS; Polysomnography
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Escitalopram
Procedure: A baseline overnight polysomnography (oPSG)

SUMMARY:
The purpose of this study is to assess the effect of escitalopram on sleep architecture utilizing a prospective design.

Hypothesis: Escitalopram will improve REM latency in patients with MDD that have responded clinically to treatment.

DETAILED DESCRIPTION:
Disturbance of sleep is a prominent symptom in depressive disorders. Alterations of sleep patterns in depressed patients include insomnia, frequent awakenings, early wake-up and non-refreshing sleep. Polysomnographic recordings have confirmed these reports, reporting reduced latency of the first REM episode of the night, with decreased density of rapid eye movements, and enhancement of total percentage of REM sleep, a reduction of deep slow wave sleep (SWS) and increase in night awakenings (Benca et al., Classification of sleep disorders).

The effects of antidepressant drugs on depression and sleep disorders, specifically SSRIs, have been thoroughly researched. The effects of escitalopram on sleep in depressed patients have been reported using a retrospective design, and in this proposed protocol, we suggest to assess the effect of escitalopram on sleep architecture utilizing a prospective design.

Hypothesis:

Escitalopram will improve REM latency in patients with MDD that have responded clinically to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from MDD, excluding a depressive episode of Bipolar Disorder.
* The depressive episode is not secondary to a general medical condition or substance abuse.
* Ages between 18-65 years old.
* Patients receiving other medications must be on a stable dosage for one month before entering the trial, including hypnotics.
* Able to understand and sign an informed consent form.

Exclusion Criteria:

* Patients suffering from sleep disturbances due to a physical condition (COPD, sleep apnea or essential insomnia preceding the diagnosis of depression).
* Patients suffering from an unstable clinically significant medical condition (cardiovascular, endocrine, nutritional, hepatic, urinary).
* Patients suffering from a malignancy or neuro-degenerative such as Parkinsons' disease
* Patients suffering from a clinically significant psychiatric psychotic disease, as judged by DSM-IV criteria, such as schizophrenia or acute psychosis.
* Patients experiencing severe withdrawal symptoms following a discontinuation of hypnotic drugs, upon entry into the baseline phase.
* History of drug or alcohol dependence within the last year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2007-02

PRIMARY OUTCOMES:
Change in latency of the first REM episode of the night.

SECONDARY OUTCOMES:
Density of rapid eye movements
Changes of total percentage of REM sleep
Changes in deep slow wave sleep (SWS)
Number of night awakenings

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Lewinski, Dr., Principal Investigator — Sheba Medical Center, Department of psychiatry; Mark Weiser, Dr., Study Chair — Sheba Medical Center, Department of psychiatry
Locations (1):
- Sheba Medical Center, Department of psychiatry, Tel Litwinsky, Israel

REFERENCES:
- [Background] Benca RM, Obermeyer WH, Thisted RA, Gillin JC. Sleep and psychiatric disorders. A meta-analysis. Arch Gen Psychiatry. 1992 Aug;49(8):651-68; discussion 669-70. doi: 10.1001/archpsyc.1992.01820080059010. PMID 1386215
- [Background] Lader M, Andersen HF, Baekdal T. The effect of escitalopram on sleep problems in depressed patients. Hum Psychopharmacol. 2005 Jul;20(5):349-54. doi: 10.1002/hup.694. PMID 15912558